CLINICAL TRIAL: NCT05019742
Title: A Double-Blind, Placebo-Controlled Trial to Investigate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of SPH3127 in Patients With Mild-to-Moderate Ulcerative Colitis
Brief Title: Evaluation of SPH3127 in Patients With Mild-to-Moderate Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Shanghai Pharma Biotherapeutics USA Inc. experienced difficulty in recruiting clinical research sites and in enrolling patients with ulcerative colitis, and consequently, the study was terminated due to futility.
Sponsor: Shanghai Pharma Biotherapeutics USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPH3127-US-01
Record Dates: First submitted 2021-08-13; First posted 2021-08-25 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis
Keywords: mild-to-moderate; selective renin inhibitor
MeSH Terms: conditions — Colitis, Ulcerative | interventions — SPH3127

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): 2 placebo tablets, 1 in the morning and 1 in the evening, daily for 8 weeks. After 8 weeks, optional randomization to 1 of 2 SPH3127 daily treatment arms for an additional 10 months
  Interventions: Drug: Placebo
- SPH3127 50 mg (Experimental): 1 50 mg SPH3127 tablet in the morning and 1 placebo tablet in the evening daily for 8 weeks.
  After 8 weeks, optional continuation of daily treatment for an additional 10 months.
  Interventions: Drug: SPH3127
- SPH3127 100 mg (Experimental): 1 50 mg SPH3127 tablet in the morning and 1 50 mg SPH3127 tablet in the evening daily for 8 weeks.
  After 8 weeks, optional continuation of daily treatment for an additional 10 months.
  Interventions: Drug: SPH3127

INTERVENTIONS:
Drug: SPH3127 — SPH3127 - selective renin inhibitor
  Arms: SPH3127 100 mg; SPH3127 50 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
SPH3127-US-01 is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, pharmacokinetics, and preliminary efficacy of SPH3127 for the treatment of mild-to-moderate ulcerative colitis.

DETAILED DESCRIPTION:
SPH3127-US-01 is a proof-of-concept multi-center, randomized, double-blind, placebo-controlled study to evaluate the safety, pharmacokinetics, and preliminary efficacy of of daily oral administration of SPH3127 or placebo for 8 weeks in patients with mild-to-moderate ulcerative colitis. After meeting all inclusion and exclusion criteria, eligible patients will be randomized to receive SPH3127 (50 mg daily, 50 mg twice daily) or placebo tablets; all patients will take 2 tablets (SPH3127 or placebo) twice a day for 8 weeks. All randomized subjects will have the opportunity to enter an active-treatment extension (50 mg SPH3127 once or twice daily) for an additional 10 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF);
2. Adult males and females ≥ 18 to < 70 years of age on the day of signing the ICF.
3. A diagnosis of UC (documented or confirmed at screening) will be eligible provided they have mild-to-moderate active UC extending ≥ 15 cm from the anal verge.
4. At screening/baseline, a Modified Mayo Clinic Score (MMCS) from 4-9, a rectal bleeding subscore ≥ 1, and a Mayo Clinic Endoscopic Subscale (MCES) score ≥ 2 determined by central reading.
5. Patient has a negative urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone) at Screening.
6. Patient has a negative alcohol breath test at Screening.
7. Female patients who have a negative pregnancy test at Screening and who agree to use adequate birth control methods throughout the entire study (and extension, if applicable) or who is post-menopausal (i.e., amenorrhea ≥ 1 year) or who have been surgically sterilized.
8. Male patients with partners of child-bearing potential who agree to use adequate birth control methods throughout the entire study (and extension, if applicable) or who have been surgically sterilized.

Exclusion Criteria:

1. Diagnosis of severe UC, defined as the presence of ≥ 6 bloody stools daily with one or more of the following: (1) oral temperature > 37.8°C or > 100.0°F; (2) pulse > 90 beats/min; (3) hemoglobin concentration < 10.5 g/dL; or erythrocyte sedimentation ratio (ESR) > 30.
2. Patients treated with oral mesalamine >2.4 g/d, systemic steroids or rectal steroids within 4 weeks prior to randomization, rectal mesalamine (within 2 weeks), immunomodulators or immunosuppressant drugs, including, but not limited to, IL-6 inhibitors, TNF inhibitors, anti-IL-1 agents and JAK inhibitors within 5 half-lives prior to randomization, antibiotics, anti-diarrheals (within 2 weeks), drugs blocking the renin-angiotensin system (e.g., direct renin inhibitors, angiotensin converting enzyme inhibitors, or angiotensin II receptor blockers) (within 4 weeks) or administration of any investigational drug (within 4 weeks). Because SPH3127 is a direct renin inhibitor with the potential to reduce blood pressure, other classes of antihypertensives (e.g., calcium channel blockers, beta blockers, diuretics, direct vasodilators, alpha blockers, central α2 antagonists) (within 4 weeks) will also be excluded. Drugs, herbal medicines and substances that inhibit or induce CYP3A4 (e.g., ritonavir, itraconazole, grapefruit juice) (within 2 weeks or 5 half-lives, whichever is longer) will be excluded.
3. History of colectomy or partial colectomy, colorectal dysplasia, Crohn's disease, toxic megacolon, or bleeding disorders.
4. A stool sample positive for enteric pathogens, including Clostridium difficile.
5. Patients with an estimated glomerular filtration rate (eGFR) < 60.
6. Patients with hepatic impairment or history of liver cirrhosis.
7. Serum creatinine > 1.5 times the upper limit of normal, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (TBIL) or alkaline phosphatase (ALP) > 2 times the upper limit of normal.
8. Serious underlying disease other than UC.
9. Previous participation in clinical trials with SPH3127
10. Known hypersensitivity to tablet ingredients or history of a significant allergic reaction to any drug as determined by the investigator.
11. Known seropositivity or positive test at screening for an active viral/bacterial infection with:

    * Hepatitis B virus (HBV) (except seropositivity due to HBV vaccination)
    * Hepatitis C virus
    * Human immunodeficiency virus
    * COVID-19 (only active infection excluded)
    * Tuberculosis
12. Known clinically relevant immunological disorders.
13. History of severe allergic or anaphylactic reactions.
14. History of malignancy, unless deemed cured by adequate treatment with no evidence of recurrence for a minimum 3 years before screening; completely eradicated non-melanoma skin cancer (such as basal cell carcinoma or squamous cell carcinoma) is not exclusionary.
15. Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g., QTcF > 450 ms or a known long QT syndrome). A first-degree heart block or sinus arrhythmia will not be considered a significant abnormality.
16. Low blood pressure at screening (i.e., SBP < 90 mmHg or DBP < 60 mmHg).
17. Clinically relevant abnormalities detected on vital signs prior to dosing.
18. Significant blood loss (including blood donation > 500 mL) or transfusion of any blood product within 12 weeks prior to the IP administration or scheduled transfusion within 4 weeks after the end of the trial.
19. Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial investigational product (IP) administration.
20. Concurrent participation, or participation within 30 days prior to the IP administration or 5 half-lives of the investigational drug (whichever is longer), in any drug/device or biologic investigational research trial.
21. Women who are breastfeeding.
22. Vaccination (including influenza and COVID-19) within the last 4 weeks prior to randomization.
23. History of drug or alcohol abuse.
24. Is an investigator, sub-investigator, research assistant, pharmacist, trial coordinator, or other staff of a relative who is directly involved in the conduct of the trial.
25. Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the trial or comply with trial procedures and requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W. Locke, PhD, Study Director — Shanghai Pharma Biotherapeutics USA Inc.
Locations (16):
- United States (16):
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Facey Medical Group at Facey Medical Foundation, Mission Hills, California
  - Precision Research Institute, San Diego, California
  - Ventura Clinical Trials, Ventura, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Velocity Clinical Research, Edgewater, Florida
  - Homestead Research Institute, Inc., Homestead, Florida
  - IHS Health, Kissimmee, Florida
  - Bayside Clinical Research LLC, Trinity, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - NY Scientific, Brooklyn, New York
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Gastro Health & Nutrition - Victoria, Victoria, Texas
  - Velocity Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients enrolled (2 placebo, 1 SPH3127 100 mg) in 16 months. Study terminated for lack of enrollment.
Pre-assignment Details: Patients must meet I/E criteria to enroll.
Groups:
- SPH3127 50 mg: 1 50 mg SPH3127 tablet in the morning and 1 placebo tablet in the evening daily for 8 weeks.
  After 8 weeks, optional continuation of daily treatment for an additional 10 months.
  SPH3127: SPH3127 - selective renin inhibitor
- SPH3127 100 mg: 1 50 mg SPH3127 tablet in the morning and 1 50 mg SPH3127 tablet in the evening daily for 8 weeks.
  After 8 weeks, optional continuation of daily treatment for an additional 10 months.
  SPH3127: SPH3127 - selective renin inhibitor
Period: Overall Study
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg
Started | 2 | 0 | 1
Completed | 2 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 3 patients enrolled, none (0) in the SPH3127 50 mg group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg | Total
Number analyzed (Participants) | 2 | 0 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 0 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Remission
Description: Number of patients with Clinical remission from baseline to Day 56
Time Frame: Screening (baseline) to Day 56
Population: No (0) subjects enrolled in SPH3127 50 mg group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg
Number analyzed (Participants) | 2 | 0 | 1
Participants | 0 | 0 | 1

2. Primary Outcome: Number of Patients With Endoscopic Remission
Description: Number of patients with Endoscopic remission from baseline to Day 56
Time Frame: Screening (baseline) to Day 56
Population: No (0) patients enrolled in SPH3127 50 mg group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg
Number analyzed (Participants) | 2 | 0 | 1
Participants | 0 | 0 | 1

3. Secondary Outcome: Number of Patients Reporting Adverse Events
Description: Number of patients reporting an adverse event (regardless of its relationship to study drug) will be tabulated and classified using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) classification system.
Time Frame: Baseline to Day 56 or date of study termination for the 3 patients (i.e., < 80 days per patient)
Population: No (0) patients enrolled in the SPH3127 50 mg group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg
Number analyzed (Participants) | 2 | 0 | 1
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 56 or date of study termination for the 3 patients (i.e., < 80 days per patient).
Description: No patients (0) enrolled in the 50 mg QD treatment group.
Arm/Group | Placebo | SPH3127 50 mg | SPH3127 100 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | SPH3127 50 mg (N=0) | SPH3127 100 mg (N=1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ulcerative colitis flare (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT05019742/Prot_SAP_001.pdf